CLINICAL TRIAL: NCT07004205
Title: The Effect of Training Based on the ARCS Motivation Model on Nursing Students' Communication Skills, Learning Motivation, and Self-Efficacy: A Randomized Controlled Trial
Brief Title: ARCS-Based Training to Improve Nursing Students' Communication, Motivation, and Self-Efficacy
Acronym: ARCS-NCOMSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Hulya Kocyigit, Research Assistant, Dr., Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Scü-Gop
Record Dates: First submitted 2025-05-12; First posted 2025-06-04 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Educational Intervention; Motivation Model
Keywords: ARCS Motivation Model; nursing students; communication skills; learning motivation; self-efficacy levels

STUDY DESIGN:
Intervention Model Description: Intervention Group Training Program (2 Weeks) Location: Classroom setting (theoretical classroom/conference hall/seminar room)
  Week 1, Day 1 (60 minutes) - Attention & Relevance
  * Introduction with background music and attention-grabbing case videos
  * Examples of nurse-patient communication (analysis of short scenarios containing communication errors)
  * Role-playing to demonstrate communication rules
  Week 1, Day 2 (60 minutes) - Confidence
  * Communication techniques (empathy, feedback, active listening)
  * In-group practices (role reversals)
  * Success-enhancing mini quizzes & positive feedback
  Week 1, Day 3 (60 minutes) - Satisfaction
  * Reward-based case analysis (small in-class rewards)
  * Participant presentations and group evaluations
  * Feedback-focused case studies
  Week 1, Day 4 (90 minutes) - Reinforcement of Entire ARCS Application
  * Scenario practice (difficult patient, emotional patient)
  * Evaluation forms & reflective journal exercises
  Week 2, Day 1 (60 minutes) - Follow-Up
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARCS (Attention, Relevance, Confidence, Satisfaction) motivation model (Experimental): ARCS (Attention, Relevance, Confidence, Satisfaction) motivation model-based training program on nursing students
  Interventions: Other: The ARCS Motivation Model Education
- Traditional Education (No Intervention): communication skills Traditional Education

INTERVENTIONS:
Other: The ARCS Motivation Model Education — The ARCS Motivation Model Education-focused on Attention, Relevance, Confidence, and Satisfaction
  Arms: ARCS (Attention, Relevance, Confidence, Satisfaction) motivation model

SUMMARY:
This study explores the impact of an ARCS-based training program on nursing students' communication skills, learning motivation, and self-efficacy. Communication is essential in nursing for quality patient care and safety, yet students often struggle with it. The ARCS Motivation Model-focused on Attention, Relevance, Confidence, and Satisfaction-aims to boost motivation and improve learning outcomes. Using a randomized controlled design, the study compares an experimental group receiving ARCS-based training with a control group receiving traditional education. Key outcomes include improved communication skills, motivation, and self-efficacy. This research highlights the potential of the ARCS model in enhancing nursing education and student performance.

DETAILED DESCRIPTION:
This study aims to examine the impact of an education program based on the ARCS Motivation Model on nursing students' communication skills, learning motivation, and self-efficacy levels. The nursing profession requires not only clinical knowledge and technical skills but also effective communication abilities, as communication plays a crucial role in enhancing patient care quality and ensuring patient safety. However, research has shown that nursing students often face deficiencies in their communication skills, which can negatively affect their professional development. Consequently, there is an increasing need for learner-centered and motivating educational approaches.

The ARCS Motivation Model, consisting of four key components-Attention, Relevance, Confidence, and Satisfaction-aims to enhance learning motivation. Literature suggests that this model positively impacts nursing students' learning processes. This study investigates whether ARCS-based training is effective in improving nursing students' communication skills, learning motivation, and self-efficacy.

The research will be conducted using a randomized controlled design with first-year nursing students from Tokat Gaziosmanpaşa University. The students will be randomly assigned to either an experimental or a control group. The experimental group will receive ARCS-based education, while the control group will receive traditional education. The study will evaluate whether there are significant differences in communication skills, learning motivation, and self-efficacy between the two groups at the end of the training process.

Data will be collected using the Effective Communication Skills Scale, Learning Motivation Scale, Self-Efficacy Scale, and a Demographic Information Form. These instruments will measure the participants' communication skills, motivation levels, and demographic characteristics. The ARCS model's four stages (Attention, Relevance, Confidence, and Satisfaction) will be applied through teaching materials and group activities during the intervention.

In conclusion, this study aims to explore the effects of an ARCS-based training model in improving nursing students' communication skills and motivation, providing insights into the effectiveness of motivation-enhancing educational methods.

ELIGIBILITY:
Inclusion Criteria

* Must be enrolled in the 1st year of the Nursing Faculty
* Must be participating in clinical practice (internship) for the first time
* Must voluntarily agree to participate in the study and sign the informed consent form
* Must agree to attend all designated sessions during the training period
* Must have proficiency in reading and writing Turkish
* Must have a suitable health condition for participation in individual and group activities

Exclusion Criteria:

Has previously participated in any clinical practice/internship

* Has previously attended specialized training on communication skills, self-efficacy, or learning motivation
* Unable to attend 2 or more sessions during the research process
* Decides to withdraw from participation during the research or withdraws consent
* Provides incomplete or incorrect responses to data (significant omissions in pre-test or post-test forms)

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
communication skills | 1 week before and 2 weeks after the intervention
  Communication Skills Measured by: Effective Communication Skills Scale (Range: 34-170; higher scores indicate better communication skills)
learning motivation | 1 week before and 2 weeks after the intervention
  MotivationMeasured by: Motivation Scale Related to Instructional Material (Range: 33-165; higher scores indicate better learning motivation)
self-efficacy levels | 1 week before and 2 weeks after the intervention
  Self-efficacy Measured by: Academic Self-Efficacy Scale (Range: 33-165; higher scores indicate better self-efficacy)

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa Universty, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I would like to share it after the research is completed.

REFERENCES:
- [Derived] Kavak HK, Kazanc S. The effect of ARCS motivational model-based education on nursing students' communication skills, learning motivation, and self-efficacy: a mixed-methods randomized controlled intervention study. BMC Med Educ. 2026 Feb 7. doi: 10.1186/s12909-026-08724-8. Online ahead of print. PMID 41654826
- See also: Related Info — https://drive.google.com/file/d/1e3KxRrzeFwGGBQP5OPoUeBG_B70u8rsJ/view?usp=sharing